CLINICAL TRIAL: NCT05066477
Title: A Randomized, Double-blind Clinical Trial Investigating the Efficacy of Salmon Bone Meal on Bone Mineral Density Among Perimenopausal Osteopenic Women
Brief Title: A Clinical Trial Investigating the Effect of Salmon Bone Meal on Bone Mass Among Osteopenic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hofseth Biocare ASA (Industry)
Collaborators: Møre og Romsdal Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CALGO-OST
Record Dates: First submitted 2021-09-22; First posted 2021-10-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2023-09

CONDITIONS: Osteopenia; Osteopenia of the Elderly
Keywords: bone meal; bone mass; bone mineral density; bone mass density; salmon bone meal
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CalGo (Salmon bone meal) (Active Comparator): 4 capsules daily of CalGo (salmon bone meal enriched with Vitamin D3) is taken per orally. Each capsule contains ~500 mg of salmon bone meal (380 mg calcium, 200 mg phosphorus, 500 mg native collagen type 2), and 10 micrograms of vitamin D3 (400 IU). Once daily dosing. Duration: 2 years.
  Interventions: Dietary Supplement: CalGo
- Maltodextrin (Placebo Comparator): 4 capsules daily of maltodextrin is taken per orally. Each capsule contains 500 mg of maltodextrin. Once daily dosing. Duration: 2 years.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: CalGo — CalGo is a natural marine collagenic bone powder from salmon. The bone powder is a 100 % microcrystalline hydroxyapatite form of calcium and phosphorus. Furthermore it contains collagen type 2 and is enriched with vitamin D3.
  Arms: CalGo (Salmon bone meal)
Other: Placebo — Pure maltodextrin
  Arms: Maltodextrin

SUMMARY:
The purpose of this study is to evaluate the efficacy of salmon bone meal in preventing bone loss among perimenopausal women with reduced bone mass density.

DETAILED DESCRIPTION:
The current study is part of a larger project called the CalGo-project. The overall purpose of the study is to use bone meal from salmon to promote skeletal health. Specifically, the effect of salmon bone meal on bone mass density among perimenopausal women (age ≥ 50 years) with osteopenia is investigated over a time period of 2 years. Salmon bone meal is composed of a natural microcrystalline hydroxyapatite form of calcium and phosphorus, collagen type 2. Past literature on mammalian sources of bone meal has indicated that this form of calcium is superior in terms of preserving bone mass density compared to traditional calcium supplements. Preserving bone mass is essential to reduce the risk of future fragility fractures. Osteopenia is a condition of reduced bone mass density and bone quality which can indicate the later onset of clinical osteoporosis. Both are conditions associated with a significant risk of fragility fractures, which are a major global health burden.

Bone mass density is measured using dual-energy X-ray absorptiometry. Markers of bone formation P1NP and CTX-1 will be measured in serum samples of participants. 100 potential participants will be screened for eligibility. Participants who meet the eligibility criteria will be randomized in a double-blind manner to receive 4 capsules daily of salmon bone meal enriched with Vitamin D3 per capsule.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* ≥ 50 years of age
* DXA T-score of > -2.5 standard deviations, but ≤ -1 (osteopenic range)
* Steady state body weight 1 month before study commencement date
* No contraindications for intake of the interventional product, including a prior diagnosis of fish allergy.
* Familiar with the Norwegian language, both in writing and orally

Exclusion Criteria:

* A diagnosis of osteoporosis (BMD T-score ≤ -2.5 SD as diagnosed by DXA), or any previously diagnosed fragility fractures on a background of osteoporosis.
* Use of drugs known to affect bone metabolism, including:

  * Glucocorticoids
  * Thyroid hormones
  * Hormone replacement therapy taken continuously for a duration of less than 6 months.
  * Long-term heparin therapy
  * Anti-convulsive drugs
  * Long-term proton pump inhibitor treatment
  * Lithium
  * Anti-osteoporotic drugs
  * Cancer therapy
  * Selective estrogen receptor modulators.
* Any disease or medical condition known to affect bone tissue, including neoplasia with or without metastasis, Paget's disease of bone, Osteomalacia, or any other disease deemed relevant by the PI.
* Gastrointestinal diseases or disturbances potentially affecting absorption of nutrients, including Crohn's disease and Celiac disease.
* Hypersensitivity to ingredients in the interventional product, including fish allergy.
* Not willing to participate in the study.
* Other reasons that the PI deems it necessary to exclude the subject.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Mean change in Bone Mass Density (BMD) of the femoral neck at Month 12, and Month 24. | Baseline, 12 Months, and 24 Months.
  Change in BMD of the femoral neck is assessed based on dual-energy X-ray absorptiometry T-scores.

SECONDARY OUTCOMES:
Mean change in Bone Mass Density (BMD) of the lumbar spine (L1-L4) at Month 12, and Month 24. | Baseline, 12 Months, and 24 Months
  Change in BMD of the lumbar spine segments L1-L4 is assessed based on dual-energy X-ray absorptiometry T-scores.
Mean change in Bone Mass Density (BMD) of the distal forearm at Month 12, and Month 24. | Baseline, 12 Months, and 24 Months
  Change in BMD of the distal forearm (distal radius) is assessed based on dual-energy X-ray absorptiometry T-scores.
Change in serum levels of markers of bone formation at Month 6, Month 12, and Month 24. | Baseline, 6 Months, 12 Months, and 24 Months.
  Serum markers of bone formation are analyzed in frozen serum samples from participants.
Change from Baseline in self-assessed quality of life on the EuroQol-5 Dimensions-3 Levels (EQ-5D-3L) instrument at Month 24. | Baseline and 24 Months
  5Q-5D-3L is a standardized instrument used to measure generic quality of life based on five distinct dimensions. EQ-5D-3L contains two parts. The first part contains five questions that the individual must answer and includes mobility (walking), self-care, usual activities, pain/discomfort, and anxiety/depression. For each item, there are three possible answers. Results are reported as a five-digit number ranging from 11111 (best health status) to 33333 (worst health status). Several methods exist for analysing these number profiles, and it is possible to convert the number profile into an index number. The second part is the EQ-VAS, where the patient self-assesses their overall health on a visual analogue scale (VAS), with 100 indicating the best health status.
Difference in number of Adverse Events between the study groups. | 3 Months, 6 Months, 12 Months, 18 Months, 24 Months
  To assess whether there is a statistically significant difference in the number of adverse events between the two study groups (CalGo [Salmon Bone Meal] and Placebo).
Difference in number of fractures between the two study groups. | 3 Months, 6 Months, 12 Months, 18 Months, 24 Months
  To assess whether there is a statistically significant difference in the number of fractures between the two study groups (CalGo [Salmon Bone Meal] and Placebo).
Difference in urine calcium in a spot urine sample between the two study groups. | Baseline, 12 Months, and 24 Months.
  Amount of calcium will be measured in spot urine samples from participants.

CONTACTS AND LOCATIONS:
Overall Officials: Øystein B Lian, MD, PhD, Principal Investigator — Møre og Romsdal Hospital Trust (Helse Møre og Romsdal), Kristiansund Hospital
Locations (3):
- Norway (3):
  - Hofseth Biocare ASA, Ålesund, Møre og Romsdal
  - Kristiansund Hospital, Kristiansund, Møre og Romsdal
  - Lovisenberg Diakonale Sykehus, Oslo

IPD SHARING:
Plan to Share IPD: No